CLINICAL TRIAL: NCT06750627
Title: Efficacy of Continuous Erector Spinae Plane Block to Reduce Postoperative Pain in Patients Undergoing Unilateral Thoracotomy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Jancolin Yani, Medical Doctor, Udayana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2708/UN14.2.2.VII.14/LT/2024
Record Dates: First submitted 2024-12-08; First posted 2024-12-27 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Continuous Erector Spinae Plane Block; Unilateral Thoracotomy
Keywords: Erector Spinae Plane Block; Unilateral Thoracotomy; Regional Anesthesia; Continuous Peripheral Nerve Block

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Continuous Erector Spinae Plane Block (Active Comparator): Participants will:
  * Undergo routine pain assessments, and recovery evaluations using tools using the Visual Analogue Scale (VAS) and Quality of Recovery-15 (QoR-15).
  * Receive continuous ESPB for analgesia with USG guidance after the surgery.
  * Receive Morphine Patient Controlled Analgesia + NSAIDs + Paracetamol
  * NSAIDs used is ketorolac, with dose of 30 mg every 8 hours
  * Paracetamol 1000 mg every 8 hours will be given
  * The PCA settings will include 30 mg of morphine diluted to 30 ml, a bolus dose of 1 ml, a lockout time of 6 minutes, 10 mg maximum dose/ 4 hours
  * Participate in follow-up visits for data collection on pain, opioid usage, and recovery quality.
  Interventions: Procedure: Continuous Erector Spinae Plane Block
- Multimodal Intravenous Analgesia (Active Comparator): Participants will:
  * Undergo routine pain assessments, and recovery evaluations using tools using the Visual Analogue Scale (VAS) and Quality of Recovery-15 (QoR-15).
  * Receive Morphine Patient Controlled Analgesia + NSAIDs + Paracetamol
  * NSAIDs used will be ketorolac of 30 mg every 8 hours
  * Paracetamol 1g every 8 hours will be given
  * The PCA settings will include 30 mg of morphine diluted to 30 ml, a bolus dose of 1 ml, a lockout time of 6 minutes, 10 mg maximum dose/ 4 hours.
  * Participate in follow-up visits for data collection on pain, opioid usage, and recovery quality.
  Interventions: Drug: Multimodal Intravenous Analgesia

INTERVENTIONS:
Procedure: Continuous Erector Spinae Plane Block — Catheter are placed between the erector spinae muscle and the transversus processus with ultrasound guidance, blocking the dorsal and ventral ramus from the thorax and abdominal spinal nerves, at the level of T5. Local anesthesia is injected. Drugs used are Bupivacaine 0.25% with volume of 25 ml.
  Other Names: ESPB
  Arms: Continuous Erector Spinae Plane Block
Drug: Multimodal Intravenous Analgesia — Multimodal intravenous analgesia refers to the use of multiple intravenous (IV) agents with different mechanisms of action to provide effective pain relief. The goal is to achieve synergistic effects that improve analgesia while minimizing the doses of individual drugs, thereby reducing side effects. This approach is often used in perioperative and acute pain management.
  Patient will receive combinations of opioid through Patient Controlled Analgesia (PCA) device, NSAIDs, and Paracetamol (Acetaminophen)
  Arms: Multimodal Intravenous Analgesia

SUMMARY:
The goal of this clinical trial is to learn if continuous Erector Spinae Plane Block (ESPB) reduces postoperative pain in patients undergoing unilateral thoracotomy. It will also evaluate the safety and effectiveness of continuous ESPB. The total participants needed will be 30 persons. The main questions it aims to answer are:

* Does continuous ESPB lower the intensity of postoperative pain compared to multimodal intravenous analgesia?
* Does continuous ESPB increase the time to first analgesic request?
* Does continuous ESPB reduce the amount of intravenous opioids required in the first 48 hours after surgery?
* Does continuous ESPB improve the overall recovery quality within 48 hours post-surgery?

Participants will:

* Receive continuous ESPB or multimodal intravenous analgesia after the surgery.
* Undergo routine pain assessments, and recovery evaluations using tools like the Visual Analogue Scale (VAS) and Quality of Recovery-15 (QoR-15).
* Participate in follow-up visits for data collection on pain, opioid usage, and recovery quality.

DETAILED DESCRIPTION:
For the Continuous ESPB Group, patients will receive continuous ESPB, NSAIDs, Paracetamol, and Morphine using Patient Controlled Analgesia (PCA) with a demand only mode.

For the Intravenous Opioid, patient will receive Non-Steroidal Anti-Inflammatory Drugs (NSAIDs), Paracetamol, and Morphine using Patient Controlled Analgesia (PCA).

ELIGIBILITY:
Inclusion Criteria:

* Patients of 21-65 years of age
* Undergoing Unilateral Thoracotomy Operation

Exclusion Criteria:

* Patients with ASA Physical Status > III
* Obese or Underweight Patients with BMI of less than 18.5 or more than 29.99
* Patients with contraindications to be given local anesthesia drugs
* Patients with contraindications to be given opioid drugs
* Patients refused to participate

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Resting Pain Score 24 hours | 24 hours
  Pain scores are recorded after 24 hours after the operation using the Visual Analogue Scale (VAS). Patients are given a scale from 0 (no pain) to 10 (worst imaginable pain). Score are measured in continuous number, and higher number represents more pain.
Resting Pain Score 48 hours | 48 hours
  Pain scores are recorded after 48 hours after the operation using the Visual Analogue Scale (VAS). Patients are given a scale from 0 (no pain) to 10 (worst imaginable pain). Score are measured in continuous number, and higher number represents more pain.
Coughing Pain Score 24 hours | 24 hours
  Coughing pain scores are recorded by asking patient to cough and evaluate their pain. Pain scores are recorded after 24 hours after the operation using the Visual Analogue Scale (VAS). Patients are given a scale from 0 (no pain) to 10 (worst imaginable pain). Score are measured in continuous number, and higher number represents more pain.
Coughing Pain Score 48 hours | 48 hours
  Coughing pain scores are recorded by asking patient to cough and evaluate their pain. Pain scores are recorded after 48 hours after the operation using the Visual Analogue Scale (VAS). Patients are given a scale from 0 (no pain) to 10 (worst imaginable pain). Score are measured in continuous number, and higher number represents more pain.

SECONDARY OUTCOMES:
Time to First Analgesia | 48 hours
  First Time to Analgesia is the time recorded since patient went out from the Recovery Room to the time the patient first pressed the demand button on the Patient Controlled Analgesia device. The time will be recorded in hours.
Opioid Consumption 24 hours | 24 hours
  Opioid consumption is the total dose that is needed by the patient during a designated time frame to achieve or maintain adequate analgesic. This will be recorded after 24 hours and 48 hours after the surgery from the Patient Controlled Analgesia device and will be expressed in Mg Morphine Equivalent (MME)
Opioid Consumption 48 hours | 48 hours
  Opioid consumption is the total dose that is needed by the patient during a designated time frame to achieve or maintain adequate analgesic. This will be recorded after 24 hours and 48 hours after the surgery from the Patient Controlled Analgesia device and will be expressed in Mg Morphine Equivalent (MME)
Quality of Recovery Preoperative | At enrollment
  Quality of Recovery is measured using the Quality of Recovery 15 (QoR-15) Questionnaire which evaluate the condition and experience of the patients. This data will be expressed in quantitative minimum score of 0 and maximum score of 150. Greater score means better outcome. The questionnaire will be given before the surgery.
Quality of Recovery 24 hours | 24 hours
  Quality of Recovery is measured using the Quality of Recovery 15 (QoR-15) Questionnaire which evaluate the condition and experience of the patients. This data will be expressed in quantitative minimum score of 0 and maximum score of 150. Greater score means better outcome. This questionnaire will be given 24 hours after the surgery
Quality of Recovery 48 hours | 48 hours
  Quality of Recovery is measured using the Quality of Recovery 15 (QoR-15) Questionnaire which evaluate the condition and experience of the patients. This data will be expressed in quantitative minimum score of 0 and maximum score of 150. Greater score means better outcome. The questionnaire will be given 48 hours after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tjokorda Gde Agung Senapathi, Professor, Study Director — Udayana University
Locations (1):
- RSUP Prof. dr. I.G.N.G. Ngoerah, Denpasar, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
The data will be deidentified and maybe shared through the author's email after there are formal request through the principal investigator email. The request must contain the intentions for the use of the data (example: for Meta-Analysis purpose)

REFERENCES:
- [Background] Moorthy A, Ni Eochagain A, Dempsey E, Wall V, Marsh H, Murphy T, Fitzmaurice GJ, Naughton RA, Buggy DJ. Postoperative recovery with continuous erector spinae plane block or video-assisted paravertebral block after minimally invasive thoracic surgery: a prospective, randomised controlled trial. Br J Anaesth. 2023 Jan;130(1):e137-e147. doi: 10.1016/j.bja.2022.07.051. Epub 2022 Sep 13. PMID 36109206
- [Background] Mehta S, Jen TTH, Hamilton DL. Regional analgesia for acute pain relief after open thoracotomy and video-assisted thoracoscopic surgery. BJA Educ. 2023 Aug;23(8):295-303. doi: 10.1016/j.bjae.2023.05.001. Epub 2023 Jun 22. No abstract available. PMID 37465231
- [Background] Koo CH, Lee HT, Na HS, Ryu JH, Shin HJ. Efficacy of Erector Spinae Plane Block for Analgesia in Thoracic Surgery: A Systematic Review and Meta-Analysis. J Cardiothorac Vasc Anesth. 2022 May;36(5):1387-1395. doi: 10.1053/j.jvca.2021.06.029. Epub 2021 Jun 29. PMID 34301447
- [Background] Ivanusic J, Konishi Y, Barrington MJ. A Cadaveric Study Investigating the Mechanism of Action of Erector Spinae Blockade. Reg Anesth Pain Med. 2018 Aug;43(6):567-571. doi: 10.1097/AAP.0000000000000789. PMID 29746445
- [Background] Gupta R, Van de Ven T, Pyati S. Post-Thoracotomy Pain: Current Strategies for Prevention and Treatment. Drugs. 2020 Nov;80(16):1677-1684. doi: 10.1007/s40265-020-01390-0. PMID 32876936
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Fawzi Hanna, M.E., Abdel Latif, S.A.M., Hussien Maamoon, R.M., Abdel-Mouty Taher, I.A.-A., 2024. Erector Spinae Plane Block for Postoperative Analgesia after Video-Assisted Thoracoscopic Surgery (VATS). QJM: An International Journal of Medicine 117, hcae070.062. https://doi.org/10.1093/qjmed/hcae070.062
- [Background] De Cassai A, Bonvicini D, Correale C, Sandei L, Tulgar S, Tonetti T. Erector spinae plane block: a systematic qualitative review. Minerva Anestesiol. 2019 Mar;85(3):308-319. doi: 10.23736/S0375-9393.18.13341-4. Epub 2019 Jan 4. PMID 30621377
- [Background] Yang HM, Choi YJ, Kwon HJ, O J, Cho TH, Kim SH. Comparison of injectate spread and nerve involvement between retrolaminar and erector spinae plane blocks in the thoracic region: a cadaveric study. Anaesthesia. 2018 Oct;73(10):1244-1250. doi: 10.1111/anae.14408. Epub 2018 Aug 16. PMID 30113699
- [Background] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Background] Chiarotto A, Maxwell LJ, Ostelo RW, Boers M, Tugwell P, Terwee CB. Measurement Properties of Visual Analogue Scale, Numeric Rating Scale, and Pain Severity Subscale of the Brief Pain Inventory in Patients With Low Back Pain: A Systematic Review. J Pain. 2019 Mar;20(3):245-263. doi: 10.1016/j.jpain.2018.07.009. Epub 2018 Aug 10. PMID 30099210
- [Background] Briscoe JB, Caso R. Pain control after thoracic surgery begins in the operating room. J Thorac Dis. 2022 Aug;14(8):2745-2747. doi: 10.21037/jtd-22-968. No abstract available. PMID 36071777
- [Background] Cao C, Zhu ZH, Yan TD, Wang Q, Jiang G, Liu L, Liu D, Wang Z, Shao W, Black D, Zhao Q, He J. Video-assisted thoracic surgery versus open thoracotomy for non-small-cell lung cancer: a propensity score analysis based on a multi-institutional registry. Eur J Cardiothorac Surg. 2013 Nov;44(5):849-54. doi: 10.1093/ejcts/ezt406. Epub 2013 Aug 15. PMID 23956268